CLINICAL TRIAL: NCT03420859
Title: The Microbiome of Infertile Couples and Its Effect on Their Reproductive Outcomes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peter Humaidan (Other)
Collaborators: Rigshospitalet, Denmark (Other); Statens Serum Institut (Other); Stork Fertility Clinic, VivaNeo, Copenhagen (Unknown); Hvidovre Fertility Clinic, Copenhagen (Unknown); Køge Fertility Clinic, Denmark (Unknown)
Responsible Party: Sponsor-Investigator, Peter Humaidan, Professor, Consultant, Regionshospitalet Viborg, Skive
Organization: Regionshospitalet Viborg, Skive (Other)
Other Study IDs: 1-16-02-404-16 (datatilsynet)
Record Dates: First submitted 2018-01-01; First posted 2018-02-05 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Abnormal Vaginal Microbiota; Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Vaginal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: qPCR for abnormal vaginal microbiota — qPCR for A.vaginae and/or G.vaginalis as developed in the pilot study (Hum Reprod. 2016 Apr;31(4):795-803. doi: 10.1093/humrep/dew026. Epub 2016 Feb 23.)

SUMMARY:
A prospective cohort study in IVF patients at 5 IVF centres in Denmark. The primary aim is to include patients positive for abnormal vaginal microbiota to an RCT (EUDRACT 2016-002385-31). Secondary aims are the prevalence of abnormal vaginal microbiota in women undergoing IVF treatment, intimate hygiene and relations to the vaginal microbiota, basic fertility work up in relation to vaginal microbiota.

DETAILED DESCRIPTION:
At the time of the interim stage of the RCT (EUDRACT 2016-002385-31), we plan to make a first cross-sectional investigation of the intimate hygiene questionnaire at baseline as compared to abnormal vaginal microbiota. We plan to make focused interview of N=30 patients to cover any additional female hygiene details not covered in the original questionnaire. After this investigation we may include new questions after the interim analysis - given that the study proceeds. In this case we plan to publish the first results of the intimate hygiene habits of the patients enrolled until interim stage.

ELIGIBILITY:
Inclusion Criteria:

* First, second or third IVF stimulation cycle at the involved clinic.
* BMI<35.
* Written informed consent.
* 18-42 years old

Exclusion Criteria:

* HIV, Hepatitis B or C positivity.
* Intrauterine malformations (Vaginal ultrasound)
* Hysterosalpinx
* Known severe renal or hepatic impairment.
* HPV CIN 2 or higher.
* Patients treated with vitamin K antagonists (warfarin)
* Known or suspected hypersensitivity to clindamycin or any other antibiotic.
* Myastenia Gravis
* Former or current inflammatory bowel disease, including Mb. Crohn and Colitis ulcerosa
* Any uncontrolled concomitant disease (e.g. uncontrolled diabetes, uncontrolled hypertension etc.)

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women fulfilling the abovementioned criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1850 (Estimated)
Dates: Start 2017-12-04 (Actual); Primary Completion 2023-08-08 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Abnormal vaginal microbiota | minimum 2-7 days from vaginal swab.
  qPCR positive diagnosis as described in intervention.

SECONDARY OUTCOMES:
Intimate hygiene | 2-5 weeks from baseline to embryo transfer
  questionnaire
Male/partner seminal microbiome | 2-4 weeks from baseline to oocyte pick-up
  DNA sequencing of seminal samples
Number of participants with Clinical pregnancy as measured by heartbeat | 7-9 weeks after inclusion.
  Tested by ultrasound scanning in week 7-9.
Number of participants achieving Live birth (defined as birth of a living child later than 23 weeks) | 36-42 weeks after inclusion
  Tested by self-reported schemes mailed to the clinics.
Cumulative live birth rate | 9 months - 24 months after inclusion
  The number of live births originating from one controlled ovarian stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Humaidan, Professor, Principal Investigator — The Fertility Clinic Skive
Locations (1):
- Fertility Clinic Skive, Skive Regional Hospital, Skive, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
By Danish law, we cannot share individual data. But pseudomized data might be available from the National Danish archives. We aim to publish as fully as possible by Danish data protection law.